CLINICAL TRIAL: NCT05891652
Title: The Effects of Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) on Postoperative Pain and Analgesic Consumption in Patients Undergoing Laparoscopic Cholecystectomy: a Randomized Double-blind Controlled Trial
Brief Title: Analgesic Effect of M-TAPA on LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Assisstant Professore, Cumhuriyet University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-TAPA on LC
Record Dates: First submitted 2023-05-16; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Post Operative Pain
Keywords: modified thoracoabdominal nerve block through perichondrial approach; postoperative pain; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: There were two randomized groups: Group M-TAPA (n=21) and Group Control (no block) (n=21). All patients had standard general anesthesia. Group M-TAPA patients had bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery. Group Control had only tramadol for posteperative pain.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blocked (Active Comparator): Patients had bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery for postoperative pain control.
  Interventions: Procedure: modified thoracoabdominal nerve block through perichondrial approach
- Control (No Intervention): Patients did not have any block or infiltration anesthesia for their postoperative pain. They only received intravenous opioid analgesic (tramadol).

INTERVENTIONS:
Procedure: modified thoracoabdominal nerve block through perichondrial approach — Following sterile conditions for bilateral M-TAPA block application, the transducer was inserted on the chondrium in the sagittal plane at the 9-10th rib level. Subsequently, a deep angle was created with the probe for visualization of the underside of the costochondrium. The sonovisible needle tip was placed just below the chondrium and saline (5 ml) was injected for site confirmation. After the confirmation, 20 ml of 0.25% bupivacaine was administered for each group for a total of 40 ml of local anesthetic. Blocks were applied using an 80 mm sonovisible needle with a 6-10 MHz linear probe under the guidance of a portable ultrasound. Same procedure applied to the contralateral side.
  Arms: Blocked

SUMMARY:
Objective: To investigate the postoperative analgesic efficacy of M-TAPA block and its effect on opioid consumption in patients undergoing laparoscopic cholecystectomy (LC) surgery.

Place and Duration of Study: Department of Anesthesiology and Reanimaton, Sivas Cumhuriyet University, Sivas, Turkey, from April 2023 to May 2023.

Methodology: There were two randomized groups: Group M-TAPA (n=21) and Group Control (no block) (n=21). All patients had standard general anesthesia. Group M-TAPA patients had bilateral M-TAPA block with 0.25% bupivacaine (total volume of 40 ml) at the end of the surgery. Group Control had only tramadol for posteperative pain. Numerical rating scale (NRS) and visual analogue scale (VAS) were used to assess postoperative pain. Total tramadol consumption was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent elective laparoscopic cholecystectomy under general anesthesia and were American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients undergoing open surgery,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 19 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
numerical rating scale scores | postoperative 24 hours
  numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
total tramadol consumption | postoperative 24 hours
  postoperative analgesic need

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
23/09/2023